CLINICAL TRIAL: NCT06956326
Title: Illuminating New Paths in the Treatment of Multiple Sclerosis Relapses - Early and Specialized Rehabilitation
Acronym: MS_Early_Rehab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lars Hvid (Other)
Responsible Party: Sponsor-Investigator, Lars Hvid, Senior Researcher, PhD, Danish Multiple Sclerosis Hospitals
Organization: Danish Multiple Sclerosis Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS_Early_Rehab
Record Dates: First submitted 2025-05-01; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis
Keywords: Neurorehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive rehab (Experimental): 10 weeks of community-based physical therapy. Participants will receive two weekly supervised physical therapy session (45-60 minutes).
  The content of this exercise program and the specific exercises and exercise methods will be planned in collaboration between MS specialists from the Danish MS hospitals, the local physical therapist, and the participant.
  Interventions: Behavioral: Intensive rehab
- Usual care (Active Comparator): 10 weeks of usual care physiotherapy, normally comprised of municipal rehabilitation as well as self-administered behavior.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Intensive rehab — Frequent moderate-to-high intensity physical therapy, provided by local physiotherapists.
  Arms: Intensive rehab
Behavioral: Usual care — Usual care physiotherapy
  Arms: Usual care

SUMMARY:
The overall purpose of this project is to develop and test an infrastructure that can ensure early and specialized rehabilitation for individuals with multiple sclerosis (MS) on their path to recovery from a relapse. If this project proves successful, it can therefore help optimize clinical practice and provide a significant contribution to the treatment of relapsing-remitting sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the Danish MS Hospitals for an inpatient rehabilitation stay
* confirmed motor relapse (within the past 6 months) by a neurologist, with disability/ functional interference characterized by change in pyramidal, and/or cerebellar functional scores of 2 or higher
* completed steroid or other acute relapse treatment, if prescribed
* age over 18 years

Exclusion Criteria:

* more than 6 months since onset of motor relapse
* medical conditions or substantial cognitive impairments that hinder participation in the study (e.g. inability to perform or understand the intensive rehabilitation)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | Change from Baseline to 52 weeks
  The Expanded Disability Status Scale measures your current level of disability.
MS Functional Composite (MSFC) Score | Change from Baseline to 52 weeks
  A standardized tool used to quantify the degree of disability in patients with multiple sclerosis (MS).

SECONDARY OUTCOMES:
MS Functional Composite (MSFC) Score | Changes from Baseline to 2 weeks and 10 weeks
  A standardized tool used to quantify the degree of disability in patients with multiple sclerosis (MS).
Handgrip strength | Changes from Baseline to 2 weeks, 10 weeks, and 52 weeks
  Maximal handgrip muscle strength of both sides.
Six spot step test (SSST) | Changes from Baseline to 2 weeks, 10 weeks, and 52 weeks
  Measure of walking balance and coordination
Five times sit to stand chair rise test (5STS) | Changes from Baseline to 2 weeks, 10 weeks, and 52 weeks
  Measure of lower extremity function
Five times sit to stand chair rise test muscle power (5STS_power) | Changes from Baseline to 2 weeks, 10 weeks, and 52 weeks
  Measure of lower extremity muscle power
Patient determined disease steps (PDDS) | Changes from Baseline to 2 weeks, 10 weeks, and 52 weeks
  Patient-reported measure of mobility disability.
MS Walking Scale (MSWS) | Changes from Baseline to 2 weeks, 10 weeks, and 52 weeks
  Patient-reported measure of walking ability.
Falls Efficacy Scale International (short FES-I) | Changes from Baseline to 2 weeks, 10 weeks, and 52 weeks
  Patient-reported measure of concerns of falls (including history of falls).
Functional Assessment of MS (FAMS) | Changes from Baseline to 2 weeks, 10 weeks, and 52 weeks
  Patient-reported measure of how MS impacts quality of life.
Modified Fatigue Impact Scale (MFIS) | Changes from Baseline to 2 weeks, 10 weeks, and 52 weeks
  Patient-reported measure of fatigue.
Manual Ability Measurement (MAM36) | Changes from Baseline to 2 weeks, 10 weeks, and 52 weeks
  Patient-reported measure of hand function related to functional questions.
Treatment Satisfactory Questionnaire (TSQ) | Evaluated at 2 weeks, 10 weeks, and 52 weeks
  Patient-reported measure of treatment satisfaction.
Multiple Sclerosis Cognitive Scale (MSCS) | Changes from baseline to 2 weeks, 10 weeks, and 52 weeks
  Patient-reported measure of cognitive function.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - The Danish MS Hospitals, Haslev
  - The Danish MS Hospitals, Ry

IPD SHARING:
Plan to Share IPD: No